CLINICAL TRIAL: NCT05263323
Title: The Effect of the Training on Adaptation to Treatment Provided to Hemodialysis Patients
Brief Title: The Effect of the Training on Adaptation to Treatment Provided to Hemodialysis Patients According to the Neuman Systems Theory on Self-Esteem and Perceived Social Support
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Ayse Asli Oktay, ASSISTANT PROFESSOR, Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: KSUAYSEASLİOKTAY001
Record Dates: First submitted 2022-01-19; First posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Nursing
Keywords: Self-esteem; patient education; hemodialysis; nursing; neuman systems theory; social support
MeSH Terms: interventions — Patient Education as Topic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group - Education Group (Experimental): Stage 1; In the intervention group, at the first stage, the data were filled with the data collection tools of the intervention group.
  Stage 2; It was made two weeks after the first visit in stage 1. "Patient education according to Neuman Systems Theory" was given to the patients who participated in the study, who received hemodialysis treatment in the center determined as the intervention group. This training was applied in the form of one-on-one training by going to the homes of the patients on the day they did not go to dialysis, within the topics determined according to the theory.
  Stage 3. It was done one month after the 2nd stage. "Patient education according to Neuman Systems Theory" was repeated to the patients, and a pre-prepared education guide called "Let's Learn Hemodialysis" was distributed and a question-answer evaluation was made.
  Stage 4; It was done one month after the 3rd stage. The data of the intervention group were collected again with data collection tools.
  Interventions: Other: Patient education
- Control Group (Active Comparator): Data collection for individuals in the control group included two stages, one at the beginning and one at the end of the study.
  The first stage was applied to the experimental group during the first stage. The data of the control group were collected with data collection tools.
  The second stage was given to the experimental group during the fourth stage. In this visit, The data of the control group were collected again with data collection tools.
  Interventions: Other: Data Collecting, No Education

INTERVENTIONS:
Other: Patient education — Providing patient education to hemodialysis patients according to Neuman Systems Model by the researcher.
  Arms: Experimental Group - Education Group
Other: Data Collecting, No Education — Data were collected at the beginning and end of the study without training the control group.
  Arms: Control Group

SUMMARY:
ABSTRACT The Effect of the Training on Adaptation to Treatment Provided to Hemodialysis Patients According to the Neuman Systems Theory on Self-Esteem and Perceived Social Support Aim: The present study was conducted to determine the effect of the training provided to hemodialysis patients according to Neuman Systems Theory on self-esteem and perceived social support in pretest-posttest comparison semi-experimental fashion.

Material and Method: The study population consisted of 108 individuals. The sampling consisted of 84 subjects, 42 of whom constituted the Study Group and 42 of whom constituted the Control Group. The study was conducted in two dialysis centers between 15.04.2017 and 15.10.2017. In the study, the data were collected with Patient Identification Form, Neuman Systems Evaluation Form, Coopersmith Self-Esteem Inventory, Social Support Perceived from Family and Friends Scale and Hemodialysis Stressor Scale. In the Study Group, the training was repeated to the individuals with the training book "Let Us Learn Hemodialysis", which was prepared by the researcher, after the one-to-one training in houses in line with the Neuman Systems Model. SPSS 20 program was used to evaluate the data. Descriptive statistical methods (number, percentage), chi-square test, paired t test were used to evaluate the data.

DETAILED DESCRIPTION:
Nursing care and education are of great importance in solving the existing or potential problems of individuals dependent on hemodialysis due to chronic kidney failure and in patients' adaptation to living with their diseases and treatment (Velioğlu 2012, Pektekin 2013). In this process, nurses benefit from nursing theory-based models to protect and improve the health of sick/healthy individuals, to ensure that they receive optimal care, and to accelerate their recovery process. One of these models is the Neuman Systems Model. The Neuman Systems Model, a well-being-oriented holistic approach that considers patients an open system, is a suitable model for holistic evaluation of patients and guiding nursing practices, as it includes five variables characterizing the individual, namely physiological, developmental, spiritual, psychological, and socio-cultural variables (Uysal et.al.2009). The model concretely defines the nursing activities and the areas in which the nurse provides service; facilitates the planning and implementation of the interventions, and can be used in most of the working areas of nursing (Özer and Gökçe,2015).

Patients undergoing hemodialysis treatment go to dialysis centers, get connected to hemodialysis machines, and fear death due to the illness, all of which cause them to feel lonely. Under this circumstance, the social support systems perceived by the individual come into play, and in case of deficiency, they experience difficulties in coping (Atik et.al.2015). National and international literature has proven that hemodialysis patients receive high social support from family, friends, and special people, which contributes positively to their treatment process, quality of life, social appearance anxiety, and self-esteem. (Atik et.al.2015; Alexopoulou et.al.2016; Silva et.al.2016; Theodoritsi et.al.2016; Karadağ et.al.2013) Many patients undergoing hemodialysis treatment for chronic kidney failure see the dialysis machine as an extension of their own body, consequently leading to deterioration in their self-esteem. Skin, bone, digestive system, nervous system changes, and fistulas related to uremia are factors that increase the loss of body image and self-esteem (Yılmaz,2014). Interventions to be implemented by the nurse to increase self-esteem help hemodialysis patients to use problem-focused coping strategies. Accordingly, improving the role of nurses in boosting patients' self-esteem increases patients' adherence to treatment and enables them to cope with problems more easily (Rezaei and Salehi,2016). National and international studies show that hemodialysis patients' beliefs about their disease and treatment play a significant role in their autonomy and self-esteem, education to improve quality of life affects/increases patients' self-esteem, hemodialysis patients with high self-esteem use problem-focused coping strategies, and individuals receiving hemodialysis treatment have lower self-esteem levels than healthy individuals (Yılmaz ,2014; Soltani-Nejad and Zeighami 2018; Rezaei and Salehi,2016; Jansen et.al.2014; Theofilou 2012).

There are studies in which nursing care and case presentations are made in line with the Neuman Systems Model in our country and the international literature (Uysal et.al.2009; Özer and Gökçe 2015; Braga et.al.2018; Ahmadi and Sadeghi 2017; Luz Omaria et.al.2016; Angosta et.al.2014; Yarcheski et.al.2010; Sultan 2018; Özkan and Öztürk 2013; Mert and Barutçu 2013; Güner and Kavlak 2015; Eren and Çalışkan 2018). These studies have shown that the integration of the model into these case presentations and nursing care reflects positively on the results and serves as a holistic guide in nursing practice. The use of models in the education program that the nurses plan within the scope of their educator role increases the effectiveness of the education, and these educational interventions reflect on the patient behaviors. Neuman Systems Model, which defines the individual as an open system, is preferred for more systematic and effective patient education in hemodialysis patients as it allows the evaluation of many stressors affecting the individual during the hemodialysis treatment process. The stages and content of the education process planned to eliminate the effects of these stressors are compatible with the nursing intervention stages of the model. Accordingly, this study aims to evaluate the effect of Neuman Systems Model guided therapeutic training given to individuals receiving hemodialysis treatment on self-esteem and perceived social support.

MATERIALS AND METHODS Type of the Research This research has a pretest-posttest comparative controlled quasi-experimental design.

Place and Time of the Research The research was carried out at Kahramanmaraş Sütçü İmam University Research and Application Hospital Hemodialysis Service and Necip Fazıl City Hospital Hüsnü Öksüz Dialysis Center between 15.04.2017 and 15.10.2017.

Universe and Sample of the Research All patients registered and treated in Kahramanmaraş Sütçü İmam University Research and Application Hospital Hemodialysis Service (Experimental group) and Necip Fazıl City Hospital Hüsnü Öksüz Dialysis Center (Control group) constituted the research universe (N:108). Experimental and control groups were formed by purposive sampling. The entire universe was included in the sample without selecting a sample. The study was carried out with 84 patients, experimental (n:42) and control (n:42). Inclusion criteria for the study;

* Being over 18 years old
* Being literate
* Not being deaf
* Being able to communicate in Turkish
* Continuing hemodialysis treatment for at least 6 months
* Not receiving a medical diagnosis of psychiatric illness
* Being conscious, cooperative

Data Collection Tools Patient Information Form The patient information form used in the study consists of a total of 23 questions. It was prepared under the guidance of the relevant literature (Özdemir and Taşçı 2013; Biçer et.al.2013; Davaridolatabadi and Abdeyazdan 2016; Mutlu ve Duyan,2012,Neuman 1996, Fawcett 2001, Alligood and Tomey 2006, Horigan and Barroso 2016) and includes questions about the patient characteristics and hemodialysis treatment characteristics.

Neuman Systems Evaluation Form The form consisting of 21 questions prepared by a thorough literature review (Velioğlu 2012, Uysal et.al.2009, Özer and Gökçe 2015, Mert and Barutçu 2013, Güner and Kavlak 2015, Alligood 2014, Fawcett and Madeya 2013, Turner and Kaylor 2015, Neuman and Fawcett 2011, Neuman 1996, Fawcett and Gigliotti 2001, Alligood and Tomey 2006) allows the patients to be evaluated based on their internal, interpersonal, and external stressors, in line with Neuman's model, which refers to the patient as an open system that interacts with these stressors.

Neuman Systems Model-Based Patient Education Guidelines After the literature review, the education topics of patients receiving hemodialysis treatment were created by the researchers within the scope of primary, secondary, and tertiary prevention intervention modes outlined in the Neuman system model (Velioğlu 2012, Özer and Gökçe 2015, Arreguy-Sena et.al.2018, Karadakovan and Kaymakçı 2011). This Neuman Systems Model-based training guideline prepared for the individuals in the experimental group was published as a training booklet called "Let's Learn Hemodialysis" and distributed to the patients. At the end of the research, the training booklet was also distributed to the individuals in the control group.

Scale of Perceived Social Support from Family (PSS-FM) and Friends (PSS-FR) The study used the "Perceived Social Support from Family and Friends Scale" developed to determine the social support score perceived by the patients from their family and friends, which was adapted into Turkish by Eskin (Eskin 1993), and confirmed for validity and reliability. The scale is two independent scales, each including 20 items (Kahriman and Polat 2003).

Coopersmith Self-Esteem Inventory (Adult Form) (SEI) The "Coopersmith Self-Esteem Inventory" consisting of 25 items was used to evaluate the self-esteem level of the patients. The reliability study in our country was conducted by Turan and it was determined as a valid and reliable scale (Turan and Tufan,1987).

Hemodialysis Stressor Scale (HSS) The hemodialysis stressor scale was adapted to Turkish society by Kara (Kara 2006). Hemodialysis Stressor Scale is a five-point Likert-type scale consisting of 23 items. An increase in the score obtained from the scale indicates an increase in the perceived stress level (Kara 2006).

Data Collection First of all, the patients in the research group were informed about the purpose and importance of the study, and their written and verbal consents were obtained for voluntary participation. Data were collected from the patients in the experimental group in four stages. In the first stage, data were collected through scales and forms. In the second stage, the patients received training prepared in line with the Neuman Systems Model at their homes on a day when they did not go to the hemodialysis unit, and a printed model-based training guide was distributed. The third stage included training repetition and question-answer steps in the dialysis center. In the fourth and final stage, data were collected once again for the last time. Data collection for individuals in the control group included two stages, one at the beginning and one at the end of the study.

Data Analysis Data analysis was performed in a computer environment using SPSS 20 software. Descriptive statistical methods (number, percentage) and chi-square test were used. Parametric tests were used as the scales had normal distribution. In the comparison of quantitative data for scales with normal distribution, independent t-test was used for the difference between the two groups, paired t-test for the pre-test post-test comparative analysis in the same group, and one-way analysis of variance for the comparison of the means of more than two groups.

Ethical Aspect of the Research Following the approval of Atatürk University Faculty of Health Sciences Ethics Committee (Number: 2016/12/04, Date: 09.01.2017), written permission was obtained from the Chief Physician of KSU Research and Application Hospital and the General Secretariat of Kahramanmaraş Public Hospitals Union to conduct the research. The purpose of the study was explained to the participating patients. Verbal and written informed consent forms were obtained.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years old
* Being literate
* Not being deaf
* Being able to communicate in Turkish
* Continuing hemodialysis treatment for at least 6 months
* Not receiving a medical diagnosis of psychiatric illness
* Being conscious, cooperative

Exclusion Criteria:

* Those who cannot communicate in Turkish
* Those who do not want to participate in the research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2017-04-15 (Actual); Primary Completion 2017-07-15 (Actual); Study Completion 2017-10-15 (Actual)

PRIMARY OUTCOMES:
The increase in perceived social support from family and friends at ten weeks after training on adherence to treatment according to the Neuman systems model. | week 10
  Scale of Perceived Social Support from Family and Friends.The scale is two independent scales and each scale has 20 items. Scores range from 0-20. It is accepted that the higher the scores, the higher the perceived social support from family and friends.
Improvement of patients' self-esteem at ten weeks after training on adherence to treatment according to the Neuman systems model. | week 10
  Coopersmith Self-Esteem Inventory (Adult Form).The Coopersmith Self-Esteem Inventory (Adult Form) consists of 25 questions. The highest score to be obtained from the scale is 100, and the lowest score is 0. If the score obtained from the scale is between 10-30 points, it indicates low self-esteem, between 30-70 points moderate and between 70-100 points indicates high self-esteem.
Decreased hemodialysis stressor levels of patients in ten weeks after training on adherence to treatment according to the Neuman systems model. | week 10
  Hemodialysis Stressor Scale.The Hemodialysis Stressor Scale is a five-point Likert-type scale consisting of 29 items. Hemodialysis Stressor Scale total score is between 29 and 145. An increase in the score obtained from the scale indicates an increase in the perceived stress level.

CONTACTS AND LOCATIONS:
Locations (1):
- Kahramanmaraş Sutçu Imam University Faculty of Health Sciences, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No